CLINICAL TRIAL: NCT04591730
Title: First-time Fathers' Experiences of Childbirth in Lorraine.
Acronym: PRIMIPERE
Status: Terminated | Type: Observational
Why Stopped: Completion failure
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, AVERCENC Léonore, Midwife, PhD, Central Hospital, Nancy, France
Other Study IDs: 2020PI138
Record Dates: First submitted 2020-10-12; First posted 2020-10-19 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Fathers; First Birth
Keywords: Fathers; Childbirth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Type I maternity: Fathers who experienced a first childbirth in a type I maternity in Lorraine.
  Interventions: Other: First time father questionnaire self-administration
- Type II maternity: Fathers who experienced a first childbirth in a type II maternity in Lorraine.
  Interventions: Other: First time father questionnaire self-administration
- Type III maternity: Fathers who experienced a first childbirth in a type III maternity in Lorraine.
  Interventions: Other: First time father questionnaire self-administration

INTERVENTIONS:
Other: First time father questionnaire self-administration — The first-time father questionnaire will be self-administrated to subjects 1 month post-birth.

SUMMARY:
The primary aim of this study is to evaluate first time father's experience during childbirth in three different maternity hospitals in Lorraine.

Secondary aims of this study is to identify domains that need improvement in order to enhance fathers's experience during childbirth.

ELIGIBILITY:
Inclusion Criteria:

* First time father after a physiological pregnancy and delivery of a healthy newborn of more than 37 gestational weeks.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Father for the first time.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2022-09-19 (Actual)

PRIMARY OUTCOMES:
First-time father questionnaire score | 1 month after birth
  Minimum value of the scale = 1, maximum value = 4, higher score represent a bad experience for the father.

CONTACTS AND LOCATIONS:
Overall Officials: Leonore Avercenc, PhD, Study Director — CHRU de Nancy
Locations (1):
- Maternité du CHRU de Nancy, Nancy, Meurthe-et-Moselle, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Premberg A, Carlsson G, Hellstrom AL, Berg M. First-time fathers' experiences of childbirth--a phenomenological study. Midwifery. 2011 Dec;27(6):848-53. doi: 10.1016/j.midw.2010.09.002. Epub 2010 Oct 16. PMID 20956030
- [Result] Premberg A, Taft C, Hellstrom AL, Berg M. Father for the first time--development and validation of a questionnaire to assess fathers' experiences of first childbirth (FTFQ). BMC Pregnancy Childbirth. 2012 May 17;12:35. doi: 10.1186/1471-2393-12-35. PMID 22594834
- [Result] Capponi I, Carquillat P, Premberg A, Vendittelli F, Guittier MJ. [Translation and validation in French of the First-Time Father Questionnaire]. Gynecol Obstet Fertil. 2016 Sep;44(9):480-6. doi: 10.1016/j.gyobfe.2016.07.011. Epub 2016 Aug 24. French. PMID 27568411